CLINICAL TRIAL: NCT03062605
Title: Reducing Microbial Levels in High Caries Risk Adults
Brief Title: Reducing Bacteria That Cause Tooth Decay
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20102774
Record Dates: First submitted 2017-02-21; First posted 2017-02-23 (Actual); Results first posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Caries, Dental; Cariostatic Agents
MeSH Terms: conditions — Dental Caries | interventions — Iodine; Povidone-Iodine; Sodium Hypochlorite

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two treatment groups and continued in parallel for the three-month duration of the study.
Who Masked: Investigator
Masking Description: This was a single blind study. The participants knew which one time treatment they were receiving, but the person doing the saliva sampling and testing did not know which treatment the participant was assigned
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment(TX) (Active Comparator): . Participants were assigned randomly to one of two treatment groups and continued in parallel for the three-month duration of the study. The first treatment group (TX) rinsed with NaOCL (0.3%) for one minute followed by rinsing with iodine (10%) for one minute
  Interventions: Drug: Iodine (Betadine); Biological: NaOCL
- Control (CT) (Active Comparator): . Participants were assigned randomly to one of two treatment groups and continued in parallel for the three-month duration of the study. The control group (CT) rinsed with iodine (10%) for minute. The CT group was a positive control. Both of these treatments were done only once at the baseline. The reminder of the three-month study was to obtain saliva samples at specific times to determining microbial levels.
  Interventions: Drug: Iodine (Betadine)

INTERVENTIONS:
Drug: Iodine (Betadine)
Biological: NaOCL
  Other Names: Clorox
  Arms: Treatment(TX)

SUMMARY:
The purpose of the study is to determine the effect of a two-step mouth rinsing procedure on reducing the germs (mutans Streptococci) that cause tooth decay. We hope that the two-step mouth rinse (0.3% NaOCl followed by 10% Povidone Iodine) decreases the tooth causing germs better than the one-step mouth rinse (10% Povidone Iodine). The mouth rinse for both treatment groups is done only once at the beginning of the study after the initial saliva samples are taken, and before a detailed examination of the teeth and gums. It is hypothesized that the treatment group receiving the NaOCl and Povidone iodine will have significantly lower microbial counts than the control group (Povidone iodine) because the NaOCl will disrupt the microbial biofilm and make the Povidone iodine more effective in decreasing the microbes in the biofilm. Microbial counts are made from Salivary samples taken from participants at baseline, one week, one month, two months and three months. The samples are tested by two commercial methods for determining microbial counts. The CariScreen Test is a rapid bioluminescence assay that quantitates the total number of all of the organisms present. The CRT test requires a culture media that is specific for the two germs (S. mutans and Lactobacillus) strongly associated with tooth decay. The results of the CRT Test are read after three days of incubation.

ELIGIBILITY:
Inclusion Criteria:

* being over 20 years of age;
* having at least one obviously cavitated tooth;
* refraining from smoking, brushing the teeth and using a mouthwash the day of the bacterial sampling;
* refraining from using a commercial mouth rinse during the three months of the study;
* having any two of the following risk factors in the Caries Management by Risk Assessment (CAMBRA) protocol which qualifies as a high caries risk.

The high caries risk factors included:

* receiving fillings within the past three years;
* snacking frequently between meals;
* presenting with hyposalivation due to medication, radiation or systemic conditions;
* visual presence of heavy plaque accumulation;
* and a minimum of 20 natural teeth.

Exclusion Criteria:

* using a systemic antibiotic within the past three months;
* currently receiving dental treatment or planning to receive treatment within the next three months (emergency treatment allowed);
* being pregnant or nursing;
* any thyroid disease or sensitivity to iodine;
* the use of a commercially available mouth rinse the day of the screening examination;
* smoking, brushing the teeth and using a mouth rinse the day of the bacterial sampling;
* not being able to make morning examinations.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-05-21 (Actual); Primary Completion 2012-02-11 (Actual); Study Completion 2012-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir W. Spolsky, DMD, MPH, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brailsford SR, Byren RW, Beighton D. Evaluation of new dip slide test for the quantification of mutans streptococci from saliva. Bericht 1998.
- [Background] Caufield PW, Gibbons RJ. Suppression of Streptococcus mutans in the mouths of humans by a dental prophylaxis and topically-applied iodine. J Dent Res. 1979 Apr;58(4):1317-26. doi: 10.1177/00220345790580040301. PMID 285102
- [Background] DenBesten P, Berkowitz R. Early childhood caries: an overview with reference to our experience in California. J Calif Dent Assoc. 2003 Feb;31(2):139-43. PMID 12636318
- [Background] Dye BA, Tan S, Smith V, Lewis BG, Barker LK, Thornton-Evans G, Eke PI, Beltran-Aguilar ED, Horowitz AM, Li CH. Trends in oral health status: United States, 1988-1994 and 1999-2004. Vital Health Stat 11. 2007 Apr;(248):1-92. PMID 17633507
- [Background] Featherstone JD, Adair SM, Anderson MH, Berkowitz RJ, Bird WF, Crall JJ, Den Besten PK, Donly KJ, Glassman P, Milgrom P, Roth JR, Snow R, Stewart RE. Caries management by risk assessment: consensus statement, April 2002. J Calif Dent Assoc. 2003 Mar;31(3):257-69. No abstract available. PMID 12693825
- [Background] Hallett KB, O'Rourke PK. Oral Biofilm activity, culture testing and caries experience in school children. International Journal of Paediatric Dentistry. 2009;19(Suppl. 2):4.
- [Background] Lenox JA, Kopczyk RA. A clinical system for scoring a patient's oral hygiene performance. J Am Dent Assoc. 1973 Apr;86(4):849-52. doi: 10.14219/jada.archive.1973.0178. No abstract available. PMID 4511175
- [Background] Matsumoto Y, Sugihara N, Koseki M, Maki Y. A rapid and quantitative detection system for Streptococcus mutans in saliva using monoclonal antibodies. Caries Res. 2006;40(1):15-9. doi: 10.1159/000088900. PMID 16352875
- [Background] Pellegrini P, Sauerwein R, Finlayson T, McLeod J, Covell DA Jr, Maier T, Machida CA. Plaque retention by self-ligating vs elastomeric orthodontic brackets: quantitative comparison of oral bacteria and detection with adenosine triphosphate-driven bioluminescence. Am J Orthod Dentofacial Orthop. 2009 Apr;135(4):426.e1-9; discussion 426-7. doi: 10.1016/j.ajodo.2008.12.002. PMID 19361723
- [Background] Slots J, Jorgensen MG. Effective, safe, practical and affordable periodontal antimicrobial therapy: where are we going, and are we there yet? Periodontol 2000. 2002;28:298-312. doi: 10.1034/j.1600-0757.2002.2801123.x. PMID 12013347
- [Background] Takahashi N, Nyvad B. Caries ecology revisited: microbial dynamics and the caries process. Caries Res. 2008;42(6):409-18. doi: 10.1159/000159604. Epub 2008 Oct 3. PMID 18832827

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment(TX): Participants were assigned randomly to one of two treatment groups and continued in parallel for the three-month duration of the study. The first treatment group (TX) rinsed with NaOCL (0.3%) for one minute followed by rinsing with iodine (10%) for one minute
  Iodine (Betadine)
  NaOCL
- Control (CT): Participants were assigned randomly to one of two treatment groups and continued in parallel for the three-month duration of the study. The control group (CT) rinsed with iodine (10%) for minute.
  Iodine (Betadine)
Period: Overall Study
Arm/Group | Treatment(TX) | Control (CT)
Started | 25 | 23
Completed | 14 | 13
Not Completed | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment(TX) | Control (CT) | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age of one female in Treatment arm and one male in Control arm were unknown
  years
    number analyzed (Participants) | 24 | 22 | 46
    (all) | 40.4 (10.2) | 38.2 (6.6) | 39.4 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 10 | 5 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Microbial Levels
Description: The CRT® Bacteria (Ivoclar Vivadent) saliva sample test is done on culture media that is specific for S. mutans and Lactobacillus. After incubation for 3 days the colonies are compared to photographic standards.
Time Frame: Baseline, 12 weeks
Population: Number analyzed includes participants retained in the study for whom CRT results were available
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment(TX) | Control (CT)
Number analyzed (Participants) | 25 | 23
Participants
  Strep Mutans >10^5 at Baseline: number analyzed (Participants) | 24 | 21
  Strep Mutans >10^5 at Baseline | 11 | 7
  Lactobacillus >10^5 at Baseline: number analyzed (Participants) | 24 | 23
  Lactobacillus >10^5 at Baseline | 15 | 15
  Strep Mutans >10^5 at 12 Weeks: number analyzed (Participants) | 14 | 13
  Strep Mutans >10^5 at 12 Weeks | 2 | 5
  Lactobacillus >10^5 at 12 Weeks: number analyzed (Participants) | 14 | 13
  Lactobacillus >10^5 at 12 Weeks | 5 | 4
Statistical Analysis 1: Comparison: Treatment(TX); Strep Mutans, Baseline-12 Weeks; Test type: Other — Inequality test; p = 0.35, McNemar — Significant at p < 0.05
Statistical Analysis 2: Comparison: Control (CT); Strep Mutans, Baseline-12 Weeks; Test type: Other — Inequality test; p = 0.29, McNemar — Significant at p<0.05
Statistical Analysis 3: Comparison: Treatment(TX); Lactobacillus, Baseline-12 Weeks; Test type: Other — Inequality test; p = 0.09, McNemar — Significant at p < 0.05
Statistical Analysis 4: Comparison: Control (CT); Lactobacillus, Baseline-12 Weeks; Test type: Other — Inequality test; p = 0.13, McNemar — Significant at p < 0.05

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Treatment(TX) | Control (CT)
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes